CLINICAL TRIAL: NCT02510820
Title: The Clinical Performance of the Biofinity Contact Lens (Comfilcon A) With Two Lens Care Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-54
Record Dates: First submitted 2015-07-16; First posted 2015-07-29 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synergi / comfilcon A (Active Comparator): Participants were randomized to wear the Synergi / comfilcon A combination for one month during the cross over study.
  Interventions: Device: comfilcon A; Device: Synergi; Other: stenfilcon A
- Biotrue / comfilcon A (Active Comparator): Participants were randomized to wear the Biotrue / comfilcon A combination for one month during the cross over study.
  Interventions: Device: comfilcon A; Device: Biotrue; Other: stenfilcon A

INTERVENTIONS:
Device: comfilcon A — soft contact lens
  Other Names: Biofinity
Device: Synergi — Multipurpose solution
  Arms: Synergi / comfilcon A
Device: Biotrue — Multipurpose solution
  Arms: Biotrue / comfilcon A
Other: stenfilcon A — daily disposable contact lenses for washout period

SUMMARY:
This will be a controlled and randomized, single-masked, crossover study in which 48 subjects will use the Biofinity Contact Lens (comfilcon A) with each of the two lens care products ('solutions'), (Synergi and Biotrue Multi-purpose Solution) for one month each. Follow-up visits for each solution will take place at one week, two weeks and four weeks: with a one-week 'wash-out' period between the solutions. Key outcome measures for this study include biomicroscopic and subjective responses to the lens/solution combinations.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age and capacity to volunteer.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They agree not to participate in other clinical research for the duration of this study.
5. They have a contact lens spherical prescription between - 0.50 to - 6.00 (inclusive)
6. They have a spectacle cylindrical correction of -1.00D (Diopters) or less in each eye.
7. At dispensing, they can attain at least 0.10 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
8. They currently use silicone hydrogel soft contact lenses.
9. They are willing to comply with the wear schedule (at least 5 days per week, ≥8 hours/day).

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They have had cataract surgery.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or lactating.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
10. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, Principal Investigator — University of Manchester
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects were not dispensed the combination of multipurpose solutions.
Groups:
- Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo: Participants were randomized to wear Synergi/comfilcon A combination for one month, then cross over to the alternative Biotrue/comfilcon A combination.
- Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo: Participants were randomized to wear Biotrue/comfilcon A combination for one month, then cross over to the alternative Synergi/comfilcon A combination.
Period: First Intervention (4 Weeks)
Arm/Group | Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo | Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo
Started | 21 | 27
Completed | 21 | 26
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (1 Week)
Arm/Group | Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo | Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo | Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo
Started | 21 | 26
Completed | 20 | 26
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Participants were randomized to wear either the Synergi/comfilcon A or Biotrue/comfilcon A combination for one month, then cross over to the alternative combination.
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 51

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Hyperaemia
Description: Conjunctival hyperaemia of Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at baseline, 1 week, 2 week, and 4 week follow-up visits. Grades 0-4, 0=normal, 4=severe.
Time Frame: Baseline, 1 week, 2 weeks, 4 weeks
Population: The differences in the sample size of the results vary due to lack of subjects attending their follow-up visits, however they completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  Baseline | 0.84 (0.24) | 0.87 (0.21)
  1 week: number analyzed (Participants) | 46 | 47
  1 week | 0.87 (0.21) | 0.87 (0.22)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 0.88 (0.24) | 0.83 (0.21)
  4 weeks: number analyzed (Participants) | 44 | 45
  4 weeks | 0.90 (0.21) | 0.82 (0.17)

2. Primary Outcome: Limbal Hyperaemia
Description: Limbal hyperaemia of Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at baseline, 1 week, 2 week, and 4 week follow-up visits. Grades 0-4, 0=normal, 4=severe.
Time Frame: Baseline, 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Synergi / Comfilcon A: Participants were randomized to wear the Synergi / comfilcon A combination for one month during the cross over study.
  comfilcon A: soft contact lens Synergi: Multipurpose solution
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  Baseline | 0.73 (0.26) | 0.77 (0.22)
  1 week: number analyzed (Participants) | 46 | 47
  1 week | 0.80 (0.23) | 0.75 (0.24)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 0.73 (0.25) | 0.70 (0.26)
  4 weeks: number analyzed (Participants) | 44 | 45
  4 weeks | 0.78 (0.22) | 0.72 (0.21)

3. Primary Outcome: Corneal Staining
Description: Corneal staining of Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at baseline, 1 week, 2 week, and 4 week follow-up visits. Grades 0-4, 0=none, 4=patch.
Time Frame: Baseline, 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  Baseline | 0.30 (0.48) | 0.17 (0.34)
  1 week: number analyzed (Participants) | 46 | 47
  1 week | 0.34 (0.40) | 0.67 (0.47)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 0.38 (0.46) | 0.59 (0.54)
  4 weeks: number analyzed (Participants) | 44 | 45
  4 weeks | 0.31 (0.42) | 0.62 (0.51)

4. Primary Outcome: Papillary Conjunctivitis
Description: Papillary conjunctivitis of Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at baseline, 1 week, 2 week, and 4 week follow-up visits. Grades 0-4, 0=normal, 4=severe.
Time Frame: Baseline, 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  Baseline | 1.04 (0.22) | 1.07 (0.24)
  1 week: number analyzed (Participants) | 46 | 47
  1 week | 1.05 (0.24) | 1.04 (0.23)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 1.05 (0.26) | 1.06 (0.20)
  4 weeks: number analyzed (Participants) | 44 | 45
  4 weeks | 1.09 (0.24) | 1.06 (0.24)

5. Primary Outcome: Comfort
Description: Subjective comfort for Synergi / comfilcon A combination and Biotrue / comfilcon A combination is assessed at 1 week visit. Scale 0-100, 0=causes pain, cannot be tolerated, 100=excellent, cannot be felt.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  Comfort after insertion | 88.7 (11.4) | 83.4 (17.9)
  Comfort before removal | 76.8 (17.2) | 72.4 (22.4)
  Overall comfort | 85.6 (11.8) | 82.8 (13.9)

6. Primary Outcome: Comfort
Description: Subjective comfort for Synergi / comfilcon A combination and Biotrue / comfilcon A combination is assessed at 2 week visit. Scale 0-100, 0=causes pain, cannot be tolerated, 100=excellent, cannot be felt.
Time Frame: 2 weeks
Population: The difference in the sample size of the results vary due to lack of subjects attending their follow-up visits, however they completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 45
units on a scale
  Comfort after insertion | 87.0 (12.6) | 85.6 (14.8)
  Comfort before removal | 78.1 (19.4) | 73.9 (20.9)
  Overall comfort | 84.7 (14.9) | 83.2 (14.8)

7. Primary Outcome: Comfort
Description: Subjective comfort for Synergi / comfilcon A combination and Biotrue / comfilcon A combination is assessed at 4 week visit. Scale 0-100, 0=causes pain, cannot be tolerated, 100=excellent, cannot be felt.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 45 | 45
units on a scale
  Comfort after insertion | 88.3 (11.0) | 87.3 (15.5)
  Comfort before removal | 76.1 (21.2) | 75.0 (20.0)
  Overall comfort | 85.3 (14.3) | 84.5 (14.0)

8. Primary Outcome: Vision
Description: Subjective assessment of vision for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 1 week visit. Scale 0-100, 0=extremely poor, intolerable levels of variation in vision, 100=excellent, no variation in vision.
Time Frame: 1 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  Distance vision | 91.1 (12.7) | 92.1 (10.4)
  Variable vision | 92.1 (12.7) | 92.1 (12.4)
  Night vision: number analyzed (Participants) | 45 | 46
  Night vision | 90.4 (12.3) | 91.6 (11.2)

9. Primary Outcome: Vision
Description: Subjective assessment of vision for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 2 week visit. Scale 0-100, 0=extremely poor, intolerable levels of variation in vision, 100=excellent, no variation in vision.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 45
units on a scale
  Distance vision | 92.8 (8.7) | 91.1 (13.0)
  Variable vision | 94.3 (9.6) | 90.5 (12.3)
  Night vision: number analyzed (Participants) | 44 | 45
  Night vision | 93.2 (8.1) | 90.8 (12.7)

10. Primary Outcome: Vision
Description: Subjective assessment of vision for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 4 week visit. Scale 0-100, 0=extremely poor, intolerable levels of variation in vision, 100=excellent, no variation in vision.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 45 | 45
units on a scale
  Distance vision | 92.5 (8.8) | 92.6 (10.4)
  Variable vision | 92.6 (12.5) | 94.1 (9.5)
  Night vision: number analyzed (Participants) | 43 | 45
  Night vision | 92.1 (8.6) | 91.9 (11.5)

11. Primary Outcome: Dryness
Description: Subjective assessment of dryness for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 1 week, 2 week, and 4 week visit. Scale 0-100, 0=extremely dry 100=not dry at all.
Time Frame: 1 week, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  1 week | 82.8 (16.3) | 79.3 (20.0)
  2 weeks | 79.5 (20.5) | 80.2 (19.8)
  4 weeks | 79.9 (20.9) | 81.7 (20.3)

12. Primary Outcome: Burning/Stinging
Description: Subjective assessment of burning/stinging for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 1 week, 2 week, and 4 week visit. Scale 0-100, 0=Extreme stinging / burning, 100=No stinging / burning sensation.
Time Frame: 1 week, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  1 week | 94.3 (13.0) | 95.7 (9.4)
  2 weeks | 96.0 (8.4) | 96.8 (8.7)
  4 weeks | 94.6 (10.9) | 96.5 (9.3)

13. Primary Outcome: Ocular Redness
Description: Subjective ocular redness of Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at 1 week, 2 week, and 4 week follow-up visits. Scale 0-100, 0=extremely poor. intolerable levels of redness, 100=excellent, no redness.
Time Frame: 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  1 week | 96.0 (9.9) | 96.8 (6.4)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 95.4 (9.6) | 96.5 (8.2)
  4 weeks: number analyzed (Participants) | 45 | 45
  4 weeks | 95.5 (8.1) | 95.7 (9.9)

14. Primary Outcome: Ease of Lens Insertion
Description: Subjective assessment of insertionfor Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 1 week, 2 week, and 4 week follow-up visits. Scale 0-100, 0=unmanageable. lenses impossible to insert, 100=excellent. no problem with lens insertion.
Time Frame: 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  1 week | 90.9 (11.8) | 93.2 (8.5)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 90.8 (8.8) | 93.4 (8.9)
  4 weeks: number analyzed (Participants) | 45 | 45
  4 weeks | 91.8 (8.7) | 93.5 (8.8)

15. Primary Outcome: Ease of Lens Removal
Description: Subjective assessment of removal for Synergi / comfilcon A combination and Biotrue / comfilcon A combination was assessed at 1 week, 2 week, and 4 week follow-up visits. Scale 0-100, 0=unmanageable. lenses impossible to remove, 100=excellent. no problem with lens remove.
Time Frame: 1 week, 2 weeks, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  1 week | 91.1 (14.0) | 92.2 (11.8)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 90.7 (11.9) | 94.0 (10.5)
  4 weeks: number analyzed (Participants) | 45 | 45
  4 weeks | 91.3 (11.2) | 94.4 (8.2)

16. Primary Outcome: Ease of Use of Solution
Description: Subjective ease of use for Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at 1 week, 2 week, and 4 week follow-up visit. Scale 0-100, 0=very difficult, 100=very easy
Time Frame: 1 week, 2 weeks, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 47 | 48
units on a scale
  1 week | 87.7 (17.3) | 92.2 (11.4)
  2 weeks | 88.2 (17.5) | 93.6 (11.0)
  4 weeks | 88.7 (15.3) | 92.7 (12.6)

17. Primary Outcome: Overall Score
Description: Subjective overall scores Synergi / comfilcon A combination and Biotrue / comfilcon A combination assessed at 1 week, 2 week, and 4 week follow-up visit. Scale 0-100, 0=extremely poor, 100=excellent, highly impressed.
Time Frame: 1 week, 2 weeks, 4 weeks
Population: Data not collected as follows: 2 weeks (1 participant) and 4 weeks (1 participant - Synergi, 1 participant - Biotrue).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Synergi / Comfilcon A | Biotrue / Comfilcon A
Number analyzed (Participants) | 46 | 47
units on a scale
  1 week | 90.3 (12.6) | 90.6 (11.7)
  2 weeks: number analyzed (Participants) | 46 | 45
  2 weeks | 88.3 (15.0) | 90.7 (12.5)
  4 weeks: number analyzed (Participants) | 45 | 45
  4 weeks | 88.8 (15.4) | 91.7 (12.7)

ADVERSE EVENTS:
Groups:
- Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo: Participants were randomized to wear the Synergi / comfilcon A combination for one month during the cross over study.
  comfilcon A: soft contact lens
  Synergi: Multipurpose solution
  Biotrue: Multipurpose solution
- Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo: Participants were randomized to wear the Biotrue / comfilcon A combination for one month during the cross over study.
  comfilcon A: soft contact lens
  Biotrue: Multipurpose solution
  Synergi: Multipurpose solution
Arm/Group | Synergi/Comfilcon A Combo, Then Biotrue/Comfilcon A Combo | Biotrue/Comfilcon A Combo, Then Synergi/Comfilcon A Combo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/27
Other Adverse Events (participants affected / at risk) | 0/21 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other